CLINICAL TRIAL: NCT05028751
Title: A Phase 1b/2 Study of the Safety, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of the Selective SYK Inhibitor Lanraplenib (LANRA) in Combination With the FLT3 Inhibitor Gilteritinib, in Patients With FLT3-mutated Relapsed or Refractory AML
Brief Title: A Study to Evaluate Lanraplenib (LANRA) in Combination With Gilteritinib in Participants With FLT3-mutated Relapsed or Refractory Acute Myeloid Leukemia (AML)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Kronos Bio (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KB-LANRA- 1001; 2022-001279-15 (EudraCT Number)
Record Dates: First submitted 2021-08-25; First posted 2021-08-31 (Actual); Results first posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-07

CONDITIONS: Acute Myeloid Leukemia; Relapsed Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Lanraplenib; LANRA; Relapsed Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — gilteritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LANRA 20 mg QD + Gilteritinib 120 mg QD (Experimental): Participants received LANRA 20 mg once daily (QD) as oral tablets in consecutive 28-day cycles starting from Cycle 1 Day 1. Participants also received gilteritinib 120 mg QD as oral tablets in consecutive 28-day cycles starting from Cycle 1 Day 2. Participants received treatment until progression/relapse or lack of at least a partial remission (PR) after 6 months of study treatment, intolerance, or withdrawal from treatment by the participant or study investigator.
  Interventions: Drug: Lanraplenib; Drug: Gilteritinib
- LANRA 40 mg QD + Gilteritinib 120 mg QD (Experimental): Participants received LANRA 40 mg QD as oral tablets in consecutive 28-day cycles starting from Cycle 1 Day 1. Participants also received gilteritinib 120 mg QD as oral tablets in consecutive 28-day cycles starting from Cycle 1 Day 2. Participants received treatment until progression/relapse or lack of at least a PR after 6 months of study treatment, intolerance, or withdrawal from treatment by the participant or study investigator.
  Interventions: Drug: Lanraplenib; Drug: Gilteritinib
- LANRA 60 mg QD + Gilteritinib 120 mg QD (Experimental): Participants received LANRA 60 mg QD as oral tablets in consecutive 28-day cycles starting from Cycle 1 Day 1. Participants also received gilteritinib 120 mg QD as oral tablets in consecutive 28-day cycles starting from Cycle 1 Day 2. Participants received treatment until progression/relapse or lack of at least a PR after 6 months of study treatment, intolerance, or withdrawal from treatment by the participant or study investigator.
  Interventions: Drug: Lanraplenib; Drug: Gilteritinib
- LANRA 90 mg QD + Gilteritinib 120 mg QD (Experimental): Participants received LANRA 90 mg QD as oral tablets in consecutive 28-day cycles starting from Cycle 1 Day 1. Participants also received gilteritinib 120 mg QD as oral tablets in consecutive 28-day cycles starting from Cycle 1 Day 2. Participants received treatment until progression/relapse or lack of at least a PR after 6 months of study treatment, intolerance, or withdrawal from treatment by the participant or study investigator.
  Interventions: Drug: Lanraplenib; Drug: Gilteritinib

INTERVENTIONS:
Drug: Lanraplenib — Orally via tablets
  Other Names: LANRA
Drug: Gilteritinib — Orally via tablets
  Other Names: XOSPATA®

SUMMARY:
The primary objective of this study is to evaluate the safety of lanraplenib (LANRA) in combination with the FMS-like tyrosine kinase 3 (FLT3) inhibitor gilteritinib, in participants with relapsed or refractory (R/R) FLT3-mutated acute myeloid leukemia (AML).

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age with acute myeloid leukemia (AML) and at least 1 prior line of therapy
* FMS-like tyrosine kinase 3 (FLT3)-mutated disease documented in a local reference laboratory at the time of consideration for enrollment in the study
* Have the ability to understand the requirements and procedures of the study and sign a written informed consent form
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1 or 2
* Adequate hepatic and renal function
* Prothrombin time (PT), activated partial thromboplastin time (aPTT) and international normalized ratio (INR) ≤1.5x upper limit of normal (ULN) unless receiving therapeutic anticoagulation
* Negative serum ß-human chorionic gonadotropin (HCG) test in women of child-bearing potential (WOCBP)
* Left ventricular ejection fraction ≥50% confirmed by echocardiogram (ECHO) or multi-gated acquisition (MUGA) scan

Exclusion Criteria:

* Known central nervous system (CNS) involvement with leukemia
* Clinical signs/symptoms of leukostasis that have failed therapy including hydroxyurea and/or leukapheresis of at least 3 days duration
* Pregnant or breastfeeding women
* Active infection with hepatitis B, C or human immunodeficiency virus (HIV) infection
* Disseminated intravascular coagulation with active bleeding or signs of thrombosis
* Known active coronavirus disease 2019 (COVID-19)
* Administration of a live attenuated virus vaccine within 35 days before Cycle 1 Day 1 (C1D1)
* History of non-myeloid malignancy except for the following: adequately treated localized basal cell, or squamous cell carcinoma of the skin, or localized melanoma (with TNM stage either Tis [melanoma in-situ] or T1aN0M0) with complete resection; cervical carcinoma in situ; superficial bladder cancer; asymptomatic prostate cancer without known metastatic disease, with no requirement for therapy or requiring only hormonal therapy and with normal prostate specific antigen for > 1 year prior to start of study therapy; or any other cancer that has been in complete remission without treatment for ≥3 years prior to enrollment
* Clinically significant heart disease
* Prolongation of the long measure between Q wave and T wave in the electrocardiogram (QT) interval at baseline
* Evidence of ongoing uncontrolled systemic bacterial, fungal, or viral infection at the time of study treatment initiation
* Current (within 30 days of study enrollment) drug-induced liver injury, chronic active hepatitis, alcoholic liver disease, nonalcoholic steatohepatitis, primary biliary cholangitis with inadequate response to ursodeoxycholic acid or other health authority approved therapy, extrahepatic obstruction caused by cholelithiasis, cirrhosis of the liver, or portal hypertension
* Ongoing (within 6 weeks of study enrollment) hepatic encephalopathy
* Ongoing immunosuppressive therapy, including systemic chemotherapy for treatment of leukemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2024-04-09 (Actual); Study Completion 2024-04-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (8):
  - University of California Los Angeles (UCLA), Los Angeles, California
  - The Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Oregon Health and Science University, Portland, Oregon
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Froedtert Hospital, Milwaukee, Wisconsin
- Spain (9):
  - Hospital Universitario 12 de Octubre, Madrid, Avenida de Córdoba Sin Número
  - Hospital Germans Trias i Pujol, Barcelona, Badalona
  - MD Anderson Cancer Center Madrid, Madrid, Calle de Arturo Soria
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Institut Català d'Oncologia - Hospital Duran i Reynals (ICO L'Hospitalet), Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitari i Politècnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 24 participants were enrolled at sites in the United States and Spain.
Pre-assignment Details: A total of 35 participants were screened, of whom 24 participants were enrolled and received study treatment.
Period: Overall Study
Arm/Group | LANRA 20 mg QD + Gilteritinib 120 mg QD | LANRA 40 mg QD + Gilteritinib 120 mg QD | LANRA 60 mg QD + Gilteritinib 120 mg QD | LANRA 90 mg QD + Gilteritinib 120 mg QD
Started | 14 | 3 | 3 | 4
Completed | 0 | 0 | 0 | 0
Not Completed | 14 | 3 | 3 | 4
Not completed — Study Terminated by Sponsor | 3 | 0 | 0 | 0
Not completed — Death | 9 | 3 | 2 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Miscellaneous | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: Consisted of all participants who received ≥ 1 dose of either study drug and had at least 1 on-treatment safety-related observation.
Groups:
- LANRA 20 mg QD + Gilteritinib 120 mg QD: Participants received LANRA 20 mg QD as oral tablets in consecutive 28-day cycles starting from Cycle 1 Day 1. Participants also received gilteritinib 120 mg QD as oral tablets in consecutive 28-day cycles starting from Cycle 1 Day 2. Participants received treatment until progression/relapse or lack of at least a PR after 6 months of study treatment, intolerance, or withdrawal from treatment by the participant or study investigator.
- Total: Total of all reporting groups
Arm/Group | LANRA 20 mg QD + Gilteritinib 120 mg QD | LANRA 40 mg QD + Gilteritinib 120 mg QD | LANRA 60 mg QD + Gilteritinib 120 mg QD | LANRA 90 mg QD + Gilteritinib 120 mg QD | Total
Number analyzed (Participants) | 14 | 3 | 3 | 4 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (19.00) | 54.0 (16.82) | 70.0 (13.45) | 74.3 (3.69) | 67.5 (16.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 1 | 2 | 9
  Male | 9 | 2 | 2 | 2 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 0 | 1 | 6
  Not Hispanic or Latino | 8 | 1 | 3 | 3 | 15
  Unknown or Not Reported | 3 | 0 | 0 | 0 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 13 | 2 | 3 | 4 | 22
  Not Reported | 1 | 0 | 0 | 0 | 1
  Other | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Treatment-emergent Adverse Event (TEAE)
Description: A TEAE was any unfavorable or unintended sign, symptom, laboratory abnormality or disease (new or exacerbated) temporally associated with the use of a study drug, whether considered causally related to the study drug or not that started after the first dose of the earliest study drug through the lesser of non-protocol anti-leukemic therapy initiation or end of treatment visit.
  A serious TEAE was defined as any TEAE that:
  * Resulted in death.
  * Was life-threatening.
  * Required or prolonged a pre-existing hospitalization.
  * Resulted in disability/incapacity.
  * Was a congenital anomaly/birth defect.
  * Was considered a significant medical event by the investigator.
  TEAEs were graded for severity based on the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 as follows:
  * Grade 1 - Mild.
  * Grade 2 - Moderate.
  * Grade 3 - Severe.
  * Grade 4 - Life-threatening.
  * Grade 5 - Death related to adverse event (AE).
Time Frame: Cycle 1 Day 1 (each cycle was 28 days) to 30 days after last dose of either LANRA or gilteritinib or initiation of non-protocol antileukemic therapy, whichever was earlier (maximum duration of treatment was 183 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | LANRA 20 mg QD + Gilteritinib 120 mg QD | LANRA 40 mg QD + Gilteritinib 120 mg QD | LANRA 60 mg QD + Gilteritinib 120 mg QD | LANRA 90 mg QD + Gilteritinib 120 mg QD
Number analyzed (Participants) | 14 | 3 | 3 | 4
Participants
  TEAEs | 14 | 3 | 3 | 4
  TESAEs | 11 | 3 | 3 | 4
  Grade 3 or Grade 4 TEAEs | 12 | 3 | 2 | 3
  AEs Leading to Death (Grade 5) | 2 | 0 | 1 | 4
  TEAEs Related to LANRA | 5 | 0 | 1 | 0
  TEAEs Related to Gilteritinib | 8 | 0 | 1 | 0
  TEAEs Leading to Dose Reduction of LANRA | 0 | 0 | 0 | 0
  TEAEs Leading to Dose Reduction of Gilteritinib | 0 | 0 | 0 | 0
  TEAEs Leading to LANRA Interruption | 9 | 0 | 0 | 2
  TEAEs Leading to Gilteritinib Interruption | 9 | 0 | 0 | 2
  TEAEs Leading to Treatment Discontinuation of LANRA | 1 | 0 | 1 | 2
  TEAEs Leading to Treatment Discontinuation of Gilteritinib | 1 | 0 | 1 | 2

2. Primary Outcome: Number of Participants Who Experienced a Dose-limiting Toxicity (DLT) for LANRA
Description: A DLT was defined as any of the following occurring within the DLT assessment period:
  * A nonhematologic toxicity of Grade ≥ 3 that was at least possibly related to LANRA (with noted exceptions).
  * Any toxicity that resulted in administration of < 80% of the cumulative, Cycle 1 dose for either LANRA or gilteritinib.
  * Grade 4 neutropenia or thrombocytopenia lasting > 28 days after treatment onset that was not attributed to active acute myeloid leukemia (AML) and was at least possibly related to LANRA.
  * Any toxicity that resulted in reduction in the dose of LANRA in Cycle 1.
  DLTs were graded for severity based on the NCI-CTCAE version 5.0 as follows:
  * Grade 3 - Severe.
  * Grade 4 - Life-threatening.
Time Frame: Cycle 1 Day 1 to pre-dose Cycle 2 Day 1 (each cycle was 28 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | LANRA 20 mg QD + Gilteritinib 120 mg QD | LANRA 40 mg QD + Gilteritinib 120 mg QD | LANRA 60 mg QD + Gilteritinib 120 mg QD | LANRA 90 mg QD + Gilteritinib 120 mg QD
Number analyzed (Participants) | 14 | 3 | 3 | 4
Participants | 0 | 0 | 0 | 0

3. Primary Outcome: Maximally Tolerated Dose (MTD)/Recommended Phase 2 Dose (RP2D) of LANRA in Combination With Standard Doses of Gilteritinib
Description: The MTD/RP2D was defined as the highest dose with either 0 of 3 or no more than 1 of 6 patients with LANRA-related DLTs. All decisions regarding dose escalation including declaration of the MTD/RP2D were made by the dose-escalation committee (DEC).
Time Frame: Cycle 1 Day 1 to pre-dose Cycle 2 Day 1 (each cycle was 28 days)
Population: The study was terminated before MTD/RP2D could be determined.
Groups:
- LANRA QD + Gilteritinib 120 mg QD: Participants received LANRA QD as oral tablets in consecutive 28-day cycles starting from Cycle 1 Day 1. Participants also received gilteritinib 120 mg QD as oral tablets in consecutive 28-day cycles starting from Cycle 1 Day 2. Participants received treatment until progression/relapse or lack of at least a PR after 6 months of study treatment, intolerance, or withdrawal from treatment by the participant or study investigator.
Arm/Group | LANRA QD + Gilteritinib 120 mg QD
Number analyzed (Participants) | 0

4. Secondary Outcome: Maximal Plasma Concentration (Cmax) of LANRA
Description: Cmax was derived from plasma concentrations of LANRA using standard non-compartmental methods and actual sample times.
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 15: Pre-dose and 0.5, 1, 2, 3, 4, 6, 8 and 24 hours post-dose.
Population: Pharmacokinetic (PK) Population: Consisted of all participants with at least 1 post-dose LANRA plasma concentration with available data at each PK assessment time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LANRA 20 mg QD + Gilteritinib 120 mg QD | LANRA 40 mg QD + Gilteritinib 120 mg QD | LANRA 60 mg QD + Gilteritinib 120 mg QD | LANRA 90 mg QD + Gilteritinib 120 mg QD
Number analyzed (Participants) | 5 | 3 | 3 | 4
ng/mL
  Cycle 1 Day 1 | 148 (59.7) | 340 (277) | 441 (146) | 694 (242)
  Cycle 1 Day 15: number analyzed (Participants) | 5 | 3 | 3 | 2
  Cycle 1 Day 15 | 181 (41.3) | 298 (111) | 591 (112) | 597 (65.1)

5. Secondary Outcome: Time to Cmax (Tmax) of LANRA
Description: Tmax was derived from plasma concentrations of LANRA using standard non-compartmental methods and actual sample times.
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 15: Pre-dose and 0.5, 1, 2, 3, 4, 6, 8 and 24 hours post-dose.
Population: PK Population: Consisted of all participants with at least 1 post-dose LANRA plasma concentration with available data at each PK assessment time point.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | LANRA 20 mg QD + Gilteritinib 120 mg QD | LANRA 40 mg QD + Gilteritinib 120 mg QD | LANRA 60 mg QD + Gilteritinib 120 mg QD | LANRA 90 mg QD + Gilteritinib 120 mg QD
Number analyzed (Participants) | 5 | 3 | 3 | 4
hours
  Cycle 1 Day 1 | 2.2 (1.3) | 3.5 (2.78) | 3.33 (2.31) | 2.5 (1.29)
  Cycle 1 Day 15: number analyzed (Participants) | 5 | 3 | 3 | 2
  Cycle 1 Day 15 | 2.8 (0.837) | 2.0 (0) | 2.0 (1.0) | 3.0 (1.4)

6. Secondary Outcome: Area of the Plasma Concentration x Time Curve From Hour 0 to the Last Measurable Time Point (AUC0-last) of LANRA
Description: AUC0-last was derived from plasma concentrations of LANRA using standard non-compartmental methods and actual sample times.
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 15: Pre-dose and 0.5, 1, 2, 3, 4, 6, 8 and 24 hours post-dose.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | LANRA 20 mg QD + Gilteritinib 120 mg QD | LANRA 40 mg QD + Gilteritinib 120 mg QD | LANRA 60 mg QD + Gilteritinib 120 mg QD | LANRA 90 mg QD + Gilteritinib 120 mg QD
Number analyzed (Participants) | 5 | 3 | 3 | 4
h*ng/mL
  Cycle 1 Day 1 | 1600 (462) | 3100 (1920) | 5240 (1550) | 7700 (1520)
  Cycle 1 Day 15: number analyzed (Participants) | 5 | 3 | 3 | 2
  Cycle 1 Day 15 | 2510 (557) | 3320 (1100) | 8430 (1860) | 8490 (1360)

7. Secondary Outcome: Cmax of Gilteritinib
Description: Cmax was derived from plasma concentrations of gilteritinib using standard non-compartmental methods and actual sample times.
Time Frame: Cycle 1 Day 15: Pre-dose and 0.5, 1, 2, 3, 4, 6, 8 and 24 hours post-dose.
Population: PK Population: Consisted of all participants with at least 1 post-dose gilteritinib plasma concentration with available data at each PK assessment time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LANRA 20 mg QD + Gilteritinib 120 mg QD | LANRA 40 mg QD + Gilteritinib 120 mg QD | LANRA 60 mg QD + Gilteritinib 120 mg QD | LANRA 90 mg QD + Gilteritinib 120 mg QD
Number analyzed (Participants) | 5 | 3 | 3 | 2
ng/mL | 434 (130) | 621 (392) | 352 (198) | 326 (168)

8. Secondary Outcome: Tmax of Gilteritinib
Description: Tmax was derived from plasma concentrations of gilteritinib using standard non-compartmental methods and actual sample times.
Time Frame: Cycle 1 Day 15: Pre-dose and 0.5, 1, 2, 3, 4, 6, 8 and 24 hours post-dose.
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | LANRA 20 mg QD + Gilteritinib 120 mg QD | LANRA 40 mg QD + Gilteritinib 120 mg QD | LANRA 60 mg QD + Gilteritinib 120 mg QD | LANRA 90 mg QD + Gilteritinib 120 mg QD
Number analyzed (Participants) | 5 | 3 | 3 | 2
hours | 5.8 (2.28) | 3 (2.65) | 5 (2.65) | 5.5 (3.54)

9. Secondary Outcome: AUC0-last of Gilteritinib
Description: AUC0-last was derived from plasma concentrations of gilteritinib using standard non-compartmental methods and actual sample times.
Time Frame: Cycle 1 Day 15: Pre-dose and 0.5, 1, 2, 3, 4, 6, 8 and 24 hours post-dose.
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | LANRA 20 mg QD + Gilteritinib 120 mg QD | LANRA 40 mg QD + Gilteritinib 120 mg QD | LANRA 60 mg QD + Gilteritinib 120 mg QD | LANRA 90 mg QD + Gilteritinib 120 mg QD
Number analyzed (Participants) | 5 | 3 | 3 | 2
h*ng/mL | 8610 (2630) | 12100 (8200) | 7460 (4870) | 6390 (3060)

10. Secondary Outcome: Composite Complete Remission (cCR) Rate Per European LeukemiaNet (ELN) 2017 Criteria
Description: Percentage of participants with cCR included CR and CR with partial hematologic recovery (CRh).
  CR required all of the following, per ELN 2017 criteria:
  * Bone marrow blasts < 5 %.
  * Absence of circulating blasts and blasts with Auer rods.
  * Absence of extramedullary disease (ie, leukemia outside of bone marrow confirmed by biopsy).
  * Absolute neutrophil count > 1.0 x 10^9/L (1,000/μL).
  * Platelet count >100 x 10^9/L (100,000/μL).
  CRh required all aforementioned CR criteria except for the below:
  * Absolute neutrophil count > 0.5 x 10^9/L (500/μL) and/or;
  * Platelet count > 50 x 10^9/L (50,000/μL).
Time Frame: Cycle 1 Day 1 until occurrence of documented CR or CRh (maximum duration of follow-up was 16.1 months).
Population: Efficacy Evaluable Population: Consisted of all participants who received ≥1 dose of either study drug and completed the first protocol-specified response assessment or discontinued study treatment for toxicity or died prior to the first response assessment. Participants with no post-baseline response assessments were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LANRA 20 mg QD + Gilteritinib 120 mg QD | LANRA 40 mg QD + Gilteritinib 120 mg QD | LANRA 60 mg QD + Gilteritinib 120 mg QD | LANRA 90 mg QD + Gilteritinib 120 mg QD
Number analyzed (Participants) | 13 | 3 | 3 | 4
percentage of participants | 0 [0 to 24.7] | 0 [0 to 70.8] | 0 [0 to 70.8] | 0 [0 to 60.2]

11. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from first qualifying response (CR/CRh) until relapse or death from any cause, as assessed by study investigators.
  CR required all of the following:
  * Bone marrow blasts < 5 %.
  * Absence of circulating blasts and blasts with Auer rods.
  * Absence of extramedullary disease (ie, leukemia outside of bone marrow confirmed by biopsy).
  * Absolute neutrophil count > 1.0 x 10^9/L (1,000/μL).
  * Platelet count >100 x 10^9/L (100,000/μL).
  CRh required all aforementioned CR criteria except for the below:
  * Absolute neutrophil count > 0.5 x 10^9/L (500/μL) and/or;
  * Platelet count > 50 x 10^9/L (50,000/μL).
  Relapse was defined as the reappearance of circulating blasts or ≥ 5% blasts in the bone marrow not attributable to any other cause or reappearance of cytologically or biopsy documented extramedullary disease.
Time Frame: From first qualifying response (CR/CRh) until relapse or death from any cause (maximum duration of follow-up was 16.1 months).
Population: Efficacy Evaluable Population: Consisted of only participants who had a CR/CRh.
Arm/Group | LANRA 20 mg QD + Gilteritinib 120 mg QD | LANRA 40 mg QD + Gilteritinib 120 mg QD | LANRA 60 mg QD + Gilteritinib 120 mg QD | LANRA 90 mg QD + Gilteritinib 120 mg QD
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: Event-free Survival (EFS)
Description: EFS was defined as the time from treatment onset until treatment failure (ie, failure to achieve CR/CRh, relapse from CR/CRh, or death from any cause).
  CR required all of the following:
  * Bone marrow blasts < 5 %.
  * Absence of circulating blasts and blasts with Auer rods.
  * Absence of extramedullary disease (ie, leukemia outside of bone marrow confirmed by biopsy).
  * Absolute neutrophil count > 1.0 x 10^9/L (1,000/μL).
  * Platelet count >100 x 10^9/L (100,000/μL).
  CRh required all aforementioned CR criteria except for the below:
  * Absolute neutrophil count > 0.5 x 10^9/L (500/μL) and/or;
  * Platelet count > 50 x 10^9/L (50,000/μL).
  Relapse was defined as the reappearance of circulating blasts or ≥ 5% blasts in the bone marrow not attributable to any other cause or reappearance of cytologically or biopsy documented extramedullary disease.
Time Frame: Cycle 1 Day 1 to treatment failure (ie, failure to achieve CR or CRh, relapse from CR/CRh or death from any cause) (maximum duration of follow-up was 16.1 months).
Population: Event free survival could not be estimated as no participants had a CR/CRh.
Arm/Group | LANRA 20 mg QD + Gilteritinib 120 mg QD | LANRA 40 mg QD + Gilteritinib 120 mg QD | LANRA 60 mg QD + Gilteritinib 120 mg QD | LANRA 90 mg QD + Gilteritinib 120 mg QD
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from enrollment until death from any cause. Overall survival was estimated using Kaplan-Meier methodology.
Time Frame: Enrollment until death from any cause (maximum duration of follow-up was 16.1 months).
Population: Safety Population: Consisted of all participants who received ≥ 1 dose of either study drug and had at least 1 on-treatment safety-related observation. Participants alive at last follow-up were censored at the date of last contact.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | LANRA 20 mg QD + Gilteritinib 120 mg QD | LANRA 40 mg QD + Gilteritinib 120 mg QD | LANRA 60 mg QD + Gilteritinib 120 mg QD | LANRA 90 mg QD + Gilteritinib 120 mg QD
Number analyzed (Participants) | 14 | 3 | 3 | 4
months | 4.0 [0.9 to 10.9] | 2.6 [2.2 to NA] — Upper limit was not reached due to low number of events. | 3.7 [1.5 to NA] — Upper limit was not reached due to low number of events. | 0.5 [0.3 to NA] — Upper limit was not reached due to low number of events.

ADVERSE EVENTS:
Time Frame: Serious AEs and Other AEs: Cycle 1 Day 1 (each cycle was 28 days) to 30 days after last dose of either LANRA or gilteritinib or initiation of non-protocol antileukemic therapy, whichever was earlier (maximum duration of treatment was 183 days). All-cause mortality: Enrollment to end of study (maximum duration of follow-up was 16.1 months).
Description: Safety Population: Consisted of all participants who received ≥ 1 dose of either study drug and had at least 1 on-treatment safety-related observation.
Arm/Group | LANRA 20 mg QD + Gilteritinib 120 mg QD | LANRA 40 mg QD + Gilteritinib 120 mg QD | LANRA 60 mg QD + Gilteritinib 120 mg QD | LANRA 90 mg QD + Gilteritinib 120 mg QD
All-Cause Mortality (participants affected / at risk) | 9/14 | 3/3 | 2/3 | 4/4
Serious Adverse Events (participants affected / at risk) | 11/14 | 3/3 | 3/3 | 4/4
Other Adverse Events (participants affected / at risk) | 14/14 | 3/3 | 3/3 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LANRA 20 mg QD + Gilteritinib 120 mg QD (N=14) | LANRA 40 mg QD + Gilteritinib 120 mg QD (N=3) | LANRA 60 mg QD + Gilteritinib 120 mg QD (N=3) | LANRA 90 mg QD + Gilteritinib 120 mg QD (N=4)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia fungal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (8) | 1 (1) | 1 (2) | 1 (2)
Hyperleukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intracranial mass (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenic colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Craniofacial fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LANRA 20 mg QD + Gilteritinib 120 mg QD (N=14) | LANRA 40 mg QD + Gilteritinib 120 mg QD (N=3) | LANRA 60 mg QD + Gilteritinib 120 mg QD (N=3) | LANRA 90 mg QD + Gilteritinib 120 mg QD (N=4)
Chills (General disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (3) | 0 (0) | 2 (4) | 0 (0)
Pyrexia (General disorders) | 2 (4) | 1 (2) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (5) | 0 (0) | 2 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 0 (0) | 2 (3) | 0 (0)
White blood cell count decreased (Investigations) | 3 (8) | 0 (0) | 1 (2) | 0 (0)
Lipase increased (Investigations) | 2 (3) | 0 (0) | 1 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 2 (13) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Bilirubin conjugated increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pantoea agglomerans test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Troponin I increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Perichondritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 5 (8) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (5) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (5) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (6) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (4) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Brain injury (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical haematoma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphoria (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute graft versus host disease (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Differentiation syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
In light of the Sponsor's decision to terminate the trial at completion of Phase 1b, all analyses were restricted to results from Phase 1b participants only. Phase 2 was not enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-05-30): https://cdn.clinicaltrials.gov/large-docs/51/NCT05028751/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-15): https://cdn.clinicaltrials.gov/large-docs/51/NCT05028751/SAP_001.pdf